CLINICAL TRIAL: NCT04122261
Title: Prospective, Multicenter, Randomized, Single-blind, Parallel-controlled Clinical Trial Protocol for the Safety and Efficacy of Clinical Applications of the Endoscopic Instrument Control System
Brief Title: A Clinical Study of Chinese Domestic Surgical Robot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDWG-NST600S-CT
Record Dates: First submitted 2019-09-28; First posted 2019-10-10 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Gallstone; Cholecystitis
MeSH Terms: conditions — Gallstones; Cholecystitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): MicroHand S robotic surgery group
  Interventions: Device: the MicroHand S endoscopic instrument control system
- control group (Experimental): da Vinci robotic surgery group
  Interventions: Device: the da Vinci endoscopic instrument control system

INTERVENTIONS:
Device: the MicroHand S endoscopic instrument control system — Using the MicroHand S endoscopic instrument control system to treat gallstone or cholecystitis in minimal invasive surgery.
  Arms: experimental group
Device: the da Vinci endoscopic instrument control system — Using the da Vinci endoscopic instrument control system to treat gallstone or cholecystitis in minimal invasive surgery.
  Arms: control group

SUMMARY:
This is a prospective, multi-center, randomized, single-blind, parallel-controlled clinical trial to evaluate the safety and efficacy of the Chinese domestic endoscopic instrument control system in clinical treatment.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of the Chinese domestic endoscopic instrument control system in clinical treatment.This clinical trial is a prospective, multi-center, randomized, single-blind, parallel-controlled study. The system used in the experimental group is the endoscopic instrument control system developed by WEGO Surgical Robot Co., Ltd., and the system used in the control group is the da Vinci endoscopic instrument control system developed by Intuitive Surgical. Before patients are enrolled in this clinical study, the researchers will do a detailed screening of the subjects based on the inclusion criteria and the exclusion criteria to determine if the patients are appropriate for the clinical study. Patients who meet the conditions of the study will be required to sign an informed consent form. Then they will be randomly assigned to the experimental group or the control group. To evaluate the primary outcome measures and secondary outcome measures and to observe the incidence of organ and vascular injury. Finally, we evaluate the safety and efficacy of the test product through the comparison of the data obtained from the experimental group and the control group during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old, male or female

2 .American Society of Anesthesiologists (ASA): Level 1, Level 2 or Level 3

3. BMI 18-30Kg/m2

4. Benign gallbladder diseases such as acute or chronic cholecystitis, gallstones and polypoid lesions of gallbladder

5. Subjects or their legal representatives/guardians voluntarily participate in clinical trials and have signed informed consent form

Exclusion Criteria:

1. Participating in any other clinical trial within 30 days before signing the informed consent form
2. Pregnancy or lactation
3. With a history of epilepsy or psychosis
4. With a history of previous operations at related sites
5. Severe cardiovascular and cerebrovascular diseases with New York grade III-IV cardiac function or pulmonary insufficiency that can't tolerate the operation
6. Severe liver and kidney insufficiency such as cirrhosis and renal failure
7. Acute cholecystitis lasting for more than 72 hours, acute cholecystitis with severe complications such as cholecystitis, gangrene, perforation, etc., and gallbladder thickness thicker than 10 mm
8. Acute cholangitis, gallstone with acute pancreatitis, primary common bile duct stones, intrahepatic bile duct stones and obstructive jaundice
9. Gallbladder cancer or protuberant lesions are suspected to be cancerous
10. Severe allergic constitution and suspected or identified addicts to alcohol or drugs
11. Abdominal infection, peritonitis, diaphragmatic hernia, severe systemic infection or metastatic diseases
12. Other situations that researchers consider it inappropriate to participate in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
surgical success rate | within 24 hours after operation
  The surgical success rate is defined as the proportion of successfully operative subjects in the experimental group or the control group.

SECONDARY OUTCOMES:
The breakage rate of gallbladder | within 12 hours after operation
  The breakage rate of gallbladder is defined as the proportion of the subjects in the experimental group or the control group with specimen breakage.
Comprehensive Complication Index (CCI) | an average of 5 days after operation
  CCI is calculated using online tools provided by http://cci.assessurgery.com. Based on the Clavien-Dindo complications grade system (appendix.1), all complications and adverse events after surgical intervention are taken into consideration. The overall incidence is measured on a scale ranging from 0 (no complication) to 100 (death).
Operative time | within 12 hours after operation
  The length of time from the beginning of the operation after the robot installation to the end of the suture of the incision.
Intraoperative bleeding | within 12 hours after operation
  The total bleeding volume from the beginning of the operation to the end of the suture of the incision. It can be calculated by measuring the blood volume in the vacuum suction device and weighing the gauze after using them to wipe the bleeding.
Postoperative pain | within 24 hours after operation
  Postoperative pain is assessed by visual analogue scale (VAS) 24-26 hours after the operation, ranging from 0 (no pain) to 10 (maximum pain).
Time to first flatus | an average of 2 days after operation
  The time from the end of the operation to the subject's first flatus after surgery.
Surgeon's satisfaction | within 12 hours after operation
  After the operation, surgeons fill a questionnaire to score the flexibility, intuition and stability of the products, as well as their sense of delay and fatigue when using the products. Each question in the score ranges from 1 to 5 points and the total score is 100.
Installation time | preoperation
  The time from the power-on of the products to the end of the connection between trocars and the operative arms.
Hospital stay | an average of 5 days after operation
  The total hospital days of subjects from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Shaihong Zhu, M.D., Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang G, Yi B, Li Z, Zhu L, Hao L, Zeng Y, Zhu S. Micro-Hand Robot-Assisted Versus da Vinci Robot-Assisted Cholecystectomy: A Multi-centre, Randomized Controlled Trial. World J Surg. 2022 Nov;46(11):2632-2641. doi: 10.1007/s00268-022-06668-w. Epub 2022 Jul 20. PMID 35857076

DOCUMENTS (2):
  • Study Protocol (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04122261/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04122261/SAP_000.pdf